CLINICAL TRIAL: NCT03608163
Title: Novel Approach for the Prevention of Hypoglycemia Associated Autonomic Failure (HAAF)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study suspended for a prolonged duration due to the Pandemic. Once research resumed project was streamlined due to insufficient resources. Study was sufficiently powered to conduct analysis for 2 of the arms. Remaining Aims were never initiated.
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Meredith Hawkins, Professor of Medicine, Albert Einstein College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-9208; R01DK079974 (NIH)
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 1; Hypoglycemia; Hypoglycemia Unawareness
Keywords: diabetes; hypoglycemia; naloxone; healthy subjects; low blood sugar
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Diabetes Mellitus | interventions — Naloxone; Diazoxide

STUDY DESIGN:
Intervention Model Description: This study is a combination of model types. In phase 1 of the study, non-diabetic participants who are susceptible to hypoglycemia-associated autonomic failure (HAAF) are identified. Only participants who are susceptible to HAAF are studied in the second and third phases. Thus, continuation of subjects identified in phase one into phase two and/or three studies follows a sequential model. The second phase follows a crossover design in which subjects receive naloxone or placebo nasal sprays in a randomized, double blinded fashion. In the third phase, subjects will receive either oral diazoxide or oral placebo (for diazoxide), in combination with naloxone nasal spray or placebo (for naloxone) nasal spray in a randomized, double blinded crossover design.
Who Masked: Participant, Investigator
Masking Description: The subject and investigator will be blinded as to which intervention(s) participant is receiving first (Drug, Drug and Placebo combination, or Placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- No intervention (Susceptibility to HAAF evaluation) (No Intervention): Susceptibility to HAAF evaluation: No intervention medication will be given during episodes of hypoglycemia.
- Naloxone (Experimental): Naloxone evaluation: Intranasal naloxone (4 mg NARCAN Nasal Spray) via a nostril twice during the first hypoglycemia episode; once at the start of insulin administration and again after one hour. Intranasal naloxone (4 mg NARCAN Nasal Spray) will again be given via a nostril twice during the second period of hypoglycemia; once at the start of insulin administration and again after one hour.
  Interventions: Drug: Naloxone
- Placebo (for Naloxone) (Placebo Comparator): Naloxone evaluation: Placebo (for naloxone) nasal spray via a nostril twice during the first hypoglycemia episode; once at the start of insulin administration and again after one hour. Placebo (for naloxone) nasal spray will again be given via a nostril twice during the second period of hypoglycemia; once at the start of insulin administration and again after one hour.
  Interventions: Drug: Placebo (for Naloxone)
- Naloxone + diazoxide (Experimental): Naloxone/Diazoxide evaluation: Up to 7 mg/kg oral diazoxide 3 hours before the first hypoglycemic episode. Intranasal naloxone (4 mg NARCAN Nasal Spray) via a nostril twice during the first hypoglycemia episode; once at the start of insulin administration and again after one hour. Intranasal naloxone (4 mg NARCAN Nasal Spray) will again be given via a nostril twice during the second period of hypoglycemia; once at the start of insulin administration and again after one hour.
  Interventions: Drug: Naloxone; Drug: Diazoxide
- Diazoxide + placebo (for naloxone) (Active Comparator): Naloxone/Diazoxide evaluation: Up to 7 mg/kg oral diazoxide 3 hours before the first hypoglycemic episode. Placebo (for naloxone) nasal spray via a nostril twice during the first hypoglycemia episode; once at the start of insulin administration and again after one hour. Placebo (for naloxone) nasal spray will again be given via a nostril twice during the second period of hypoglycemia; once at the start of insulin administration and again after one hour.
  Interventions: Drug: Diazoxide; Drug: Placebo (for Naloxone)
- Naloxone + placebo (for diazoxide) (Active Comparator): Naloxone/Diazoxide evaluation: Oral placebo (for diazoxide) 3 hours before the first hypoglycemic episode. Intranasal naloxone (4 mg NARCAN Nasal Spray) via a nostril twice during the first hypoglycemia episode; once at the start of insulin administration and again after one hour. Intranasal naloxone (4 mg NARCAN Nasal Spray) will again be given via a nostril twice during the second period of hypoglycemia; once at the start of insulin administration and again after one hour.
  Interventions: Drug: Naloxone; Drug: Placebo (for Diazoxide)
- Placebo (for naloxone) + placebo (for diazoxide) (Placebo Comparator): Naloxone/Diazoxide evaluation: Oral placebo (for diazoxide) 3 hours before the first hypoglycemic episode. Placebo (for naloxone) nasal spray via a nostril twice during the first hypoglycemia episode; once at the start of insulin administration and again after one hour. Placebo (for naloxone) nasal spray will again be given via a nostril twice during the second period of hypoglycemia; once at the start of insulin administration and again after one hour.
  Interventions: Drug: Placebo (for Naloxone); Drug: Placebo (for Diazoxide)

INTERVENTIONS:
Drug: Naloxone — Naloxone Nasal Spray
  Other Names: NARCAN Nasal Spray
  Arms: Naloxone; Naloxone + diazoxide; Naloxone + placebo (for diazoxide)
Drug: Diazoxide — Diazoxide (oral)
  Arms: Diazoxide + placebo (for naloxone); Naloxone + diazoxide
Drug: Placebo (for Naloxone) — Sterile water nasal spray
  Arms: Diazoxide + placebo (for naloxone); Placebo (for Naloxone); Placebo (for naloxone) + placebo (for diazoxide)
Drug: Placebo (for Diazoxide) — Taste matched oral placebo for diazoxide
  Arms: Naloxone + placebo (for diazoxide); Placebo (for naloxone) + placebo (for diazoxide)

SUMMARY:
The overall goal of this study is to develop a new and practical way to prevent the development of Hypoglycemia Associated Autonomic Failure (HAAF), which is unawareness of hypoglycemia (low blood sugar) in individuals with diabetes. Previous studies suggest that two medications, naloxone and diazoxide, may increase the body's ability to respond to episodes of low blood sugar and prevent the development of HAAF (or hypoglycemia unawareness). Only healthy subjects are being recruited for this study. The study has three distinct phases. In the first phase, healthy, non-diabetic individuals who are susceptible to developing HAAF are identified. Only these individuals will be studied in the second and third phases. The second phase of this study evaluates the effect of using a naloxone nasal spray versus a placebo nasal spray in improving the body's response to episodes of low blood sugar and in preventing the development of HAAF. The third phase of this study evaluates the effect of using naloxone nasal spray and diazoxide in combination, compared to naloxone nasal spray plus a placebo (for diazoxide) or diazoxide plus a placebo (for naloxone) in improving the body's response to episodes of low blood sugar and in preventing the development of HAAF.

DETAILED DESCRIPTION:
Type I diabetes affects the body's ability to respond to low blood sugar (hypoglycemia). Repeated episodes of hypoglycemia may affect an individual's autonomic system, and leads to Hypoglycemia Associated Autonomic Failure (HAAF) in around two-thirds of individuals. This study is looking at healthy, non-diabetic individuals who are susceptible to developing HAAF and their response to either naloxone nasal spray alone or in combination with diazoxide in improving their body's ability to respond to episodes of low blood sugar, and in preventing the development of HAAF.

The body's response to episodes of hypoglycemia is measured using a procedure called a hypoglycemic clamp. Each phase of this study involves three clamp procedures over a period of 2 days. During the clamp procedures, glucose (a sugar) and insulin (a hormone produced in the pancreas that regulates the amount of glucose in the blood) are infused with an intravenous catheter, and blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones, including epinephrine, that are found in the body and are related to glucose metabolism. The rates of endogenous glucose production (a measure of the body's production of sugar) will be measured. Additionally, the level of awareness of hypoglycemia symptoms will be monitored using a standardized questionnaire.

Both hypoglycemia and stress activate the body's opioid system. Recently published data has shown that blocking opioid receptors with naloxone may increase the body's ability to respond to hypoglycemia.The body's response to hypoglycemia affects many systems, and acting on several of these systems may help the body to respond more effectively to episodes of low blood sugar, and to prevent the development of HAAF. Studies have shown that potassium channels in the hypothalamus, a part of the brain, have an important role in detecting hypoglycemia. Diazoxide activates potassium channels in the cells of the brain that respond to changes in sugar (glucose) that occur in the body, and may also reduce the development of hypoglycemia associated autonomic failure. Additionally, certain glucose-responsive cells in the brain have opioid receptors that are combined with potassium channels which may respond to both diazoxide and naloxone which may work together to more effectively increase the body's ability to respond to episodes of low blood sugar and prevent HAAF.

UPDATE: This study was terminated early and only the second phase (Aim 2) of the study above was conducted. This phase was designed to assess the effect of opioid receptor antagonist - intranasal naloxone - as compared to matched placebo on experimentally induced HAAF in healthy, nondiabetic volunteers.

ELIGIBILITY:
Inclusion Criteria:

-Healthy, non-diabetic subjects 21-55 years old

Exclusion Criteria:

* Body Mass Index (BMI) >35kg/m2
* If Blood Pressure (BP) >150/90 or <90/60 on repeated measurements and on more than one occasion
* Uncontrolled hyperlipidemia defined as Triglycerides >400 mg/dL and/or total cholesterol >300 mg/dL
* Clinically significant liver dysfunction: including thrombocytopenia (platelets <100,000/uL), anemia (as below), hypoalbuminemia (<3.5 g/dL), coagulopathy (INR > 1.5), and/or liver enzymes more than 3 times the upper limit of normal
* Clinically significant kidney dysfunction: Glomerular Filtration Rate (GFR): <60 mg/dL
* Clinically significant anemia: Prospective subjects with hemoglobin below the lower limit of 12 g/dL for for men and 11 g/dL for women will be assessed with history and physical exam to rule out clinically significant anemia, defined as an individual with symptoms (e.g. fatigue, weakness, shortness of breath, palpitations), signs (pallor, brittle nails etc.), or currently under treatment for anemia. In the absence of a documented hemoglobin decrease or iron deficiency, subjects will not be excluded.
* Clinically significant leukocytosis or leukopenia
* Clinically significant thrombocytopenia or thrombocytosis
* Coagulopathy
* Positive drug screen for amphetamines, barbiturates, benzodiazepines, cocaine, methadone, opiates, oxycodone, Phencyclidine (PCP). Occasional use of cannabis (not more than twice per week) is not an exclusion. If the test is read as "indeterminate" it will be repeated at the bedside and an additional sample will be sent to the lab.
* Use of medications such as beta-blockers or medications that affect counterregulatory response to hypoglycemia
* Urinalysis: clinically significant abnormalities
* Clinically significant electrolyte abnormalities
* Smoking >10 cigarettes/day
* Heavy alcohol use defined as: Men >14 drinks/week or > 4 drinks/day, Women > 7 drinks/week or > 3 drinks/day
* History of chronic liver disease, active hepatitis infection, HIV/AIDS, chronic kidney disease (stage 3 or greater), active cancer, cardiovascular disease or other heart disease, systemic rheumatologic conditions, seizures, bleeding disorders, muscle disease
* Surgeries that involve removal of endocrine glands except for thyroidectomy (if euthyroid on thyroid hormone replacement - if such history Free Thyroxine (fT4) and Thyroid Stimulating Hormone (TSH) will be checked)
* Pregnancy
* Subject enrolled in another medication intervention study less than one month prior to their anticipated start date in this study besides those done by our group
* Family history of diabetes or premature cardiac death in first degree relatives
* Allergies to medications administered during study
* Uncontrolled psychiatric disorders
* Any condition which in the opinion of the PI makes the subject ill-suited for participation in the study

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Hawkins, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 patients were consented and enrolled into Aim 2 of the study.
Groups:
- Naloxone First, Then Placebo: Naloxone evaluation: Intranasal naloxone (4 mg NARCAN Nasal Spray) via a nostril twice during the first hypoglycemia episode; once at the start of insulin administration and again after one hour. Intranasal naloxone (4 mg NARCAN Nasal Spray) will again be given via a nostril twice during the second period of hypoglycemia; once at the start of insulin administration and again after one hour.
  Naloxone: Naloxone Nasal Spray
  Placebo (for Naloxone): Sterile water nasal spray
- Placebo (for Naloxone), Then Naloxone: Naloxone evaluation: Placebo (for naloxone) nasal spray via a nostril twice during the first hypoglycemia episode; once at the start of insulin administration and again after one hour. Placebo (for naloxone) nasal spray will again be given via a nostril twice during the second period of hypoglycemia; once at the start of insulin administration and again after one hour.
  Naloxone: Naloxone Nasal Spray
  Placebo (for Naloxone): Sterile water nasal spray
Period: 1st Intervention (2 Days)
Arm/Group | Naloxone First, Then Placebo | Placebo (for Naloxone), Then Naloxone
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Washout (~6 Months)
Arm/Group | Naloxone First, Then Placebo | Placebo (for Naloxone), Then Naloxone
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: 2nd Intervention (2 Days)
Arm/Group | Naloxone First, Then Placebo | Placebo (for Naloxone), Then Naloxone
Started | 2 | 2
Completed | 2 | 1
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Naloxone evaluation: Intranasal naloxone (4 mg NARCAN Nasal Spray) via a nostril twice during the first hypoglycemia episode; once at the start of insulin administration and again after one hour. Intranasal naloxone (4 mg NARCAN Nasal Spray) will again be given via a nostril twice during the second period of hypoglycemia; once at the start of insulin administration and again after one hour.
  Naloxone evaluation: Placebo (for naloxone) nasal spray via a nostril twice during the first hypoglycemia episode; once at the start of insulin administration and again after one hour. Placebo (for naloxone) nasal spray will again be given via a nostril twice during the second period of hypoglycemia; once at the start of insulin administration and again after one hour.
  Naloxone: Naloxone Nasal Spray
  Placebo (for Naloxone): Sterile water nasal spray
Arm/Group | All Participants
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI was determined at baseline and reported in kilograms/meters-squared (kg/m^2).
  kg/m^2 | 24.9 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Peak Epinephrine Levels Between First and Third Hypoglycemic Clamp Episodes
Description: Peak epinephrine levels during the first (during Day 1) and third (During Day 2) hypoglycemic clamp episodes were compared. Blood samples were taken every 15 minutes throughout clamp procedures and analyzed using high performance liquid chromatography to measure epinephrine levels. Peak epinephrine levels during the course of the three clamp procedures over the two days were identified for each participant. Results are summarized and reported by study arm using basic descriptive statistics. A reduction of >20% in the average peak epinephrine levels between first and third hypoglycemic clamp episodes will be considered to define HAAF.
Time Frame: Obtained every 15 minutes during the first and third 2-hour hypoglycemic episodes (on Day 1 and Day 2), crossover visits up to approximately 6 months apart
Measure: Mean (Standard Error); unit: pg/mL
Groups:
- Naloxone: Naloxone evaluation: Intranasal naloxone (4 mg NARCAN Nasal Spray) via a nostril twice during the first hypoglycemia episode; once at the start of insulin administration and again after one hour. Intranasal naloxone (4 mg NARCAN Nasal Spray) will again be given via a nostril twice during the second period of hypoglycemia; once at the start of insulin administration and again after one hour.
  Naloxone: Naloxone Nasal Spray
  Placebo (for Naloxone): Sterile water nasal spray
- Placebo (for Naloxone): Naloxone evaluation: Placebo (for naloxone) nasal spray via a nostril twice during the first hypoglycemia episode; once at the start of insulin administration and again after one hour. Placebo (for naloxone) nasal spray will again be given via a nostril twice during the second period of hypoglycemia; once at the start of insulin administration and again after one hour.
  Naloxone: Naloxone Nasal Spray
  Placebo (for Naloxone): Sterile water nasal spray
Arm/Group | Naloxone | Placebo (for Naloxone)
Number analyzed (Participants) | 3 | 4
pg/mL
  1st hypoglycemic clamp episode (Day 1) | 372 (134) | 707 (195)
  3rd hypoglycemic clamp episode (Day 2) | 397 (168) | 601 (55)

2. Secondary Outcome: Endogenous Glucose Production (EGP)
Description: EGP, a measure of the body's production of sugar, was assessed by determining the Glucose Infusion Rate (GIR), an indirect measure of endogenous glucose production, during the first and third hypoglycemic clamp episodes. GIR is reported in cubic centimeters/minute (cc/min) and results are summarized and reported by study arm using basic descriptive statistics.
Time Frame: Obtained every 15 minutes during the 1st and 3rd 2-hour hypoglycemic episodes (on Day 1 and Day 2), crossover visits up to ~6 months apart. Data from the five timepoints over the final hour of the 1st and 3rd clamp episodes were averaged/reported.
Population: GIR data was obtained from 1 participant following Naloxone administration and 3 participants following Placebo administration.
Measure: Mean (Standard Error); unit: cc/min
Arm/Group | Naloxone | Placebo (for Naloxone)
Number analyzed (Participants) | 1 | 3
cc/min
  1st hypoglycemic clamp episode (Day 1) | 1.6 (NA) — Standard error is not able to be determined for the Naloxone participant due to sample size of 1. | 0.7 (0.2)
  3rd hypoglycemic clamp episode (Day 2) | 0.9 (NA) — Standard error is not able to be determined for the Naloxone participant due to sample size of 1. | 1.1 (0.3)

3. Secondary Outcome: Symptoms of Low Blood Sugar
Description: Symptoms of low blood sugar were assessed during steady state (the last 30 minutes) using the Edinburgh Hypoglycemia Symptom Scale (EHSS). The EHSS questionnaire is comprised 11 key symptoms (sweating, palpitations, shaking, hunger, confusion, drowsiness, odd behavior, speech difficulty, incoordination, nausea, and headache) and asked participants to evaluate these symptoms using an 8-point Likert scale ranging from 0 ("Not at all") to 7 ("Very severe"), for an overall possible range of 0-77 for each patient, such that higher scores are associated with more intense hypoglycemic symptoms. EHSS scores were summed and averaged and reported by study arm using basic descriptive statistics.
Time Frame: as for outcome 1
Population: Symptoms of low blood sugar scores were able to be collected from 1 participant following Naloxone administration and 3 participants following Placebo administration.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Naloxone | Placebo (for Naloxone)
Number analyzed (Participants) | 1 | 3
score on a scale
  1st hypoglycemic clamp episode (Day 1) | 2.0 (NA) — Standard error is not able to be determined for the Naloxone participant due to sample size of 1. | 4.5 (2.1)
  3rd hypoglycemic clamp episode (Day 2) | 1.2 (NA) — Standard error is not able to be determined for the Naloxone participant due to sample size of 1. | 4.2 (2.4)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed on two consecutive days over two series of visits scheduled up to approximately 6 months apart.
Description: For purposes of this study any of the 11 key symptoms assessed as part of the Edinburgh Hypoglycemia Symptom Scale were not considered adverse events unless glucose levels fell below the safe target level of 53 mg/dL, or medical attention for hypoglycemia was required. Based on this definition, none of the 4 participants in this study experienced either a Serious Adverse Event or Other (Not Including Serious) Adverse Events (AEs).
Arm/Group | Naloxone | Placebo (for Naloxone)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT03608163/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT03608163/ICF_001.pdf